CLINICAL TRIAL: NCT00014807
Title: Reducing Pesticide Exposure in Minority Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Purpose: Prevention
Other Study IDs: 8707-CP-001
Record Dates: First submitted 2001-04-11; First posted 2001-04-12 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Disorders of Environmental Origin
Keywords: Pesticide exposure; Organophosphate; Biomarkers of exposure; Poisoning; Occupational Health
MeSH Terms: conditions — Disorders of Environmental Origin; Poisoning

INTERVENTIONS:
Behavioral: Reducing Pesticide Exposure in Minority Families

SUMMARY:
This is a community-based participatory research program focusing on pesticide contamination in migrant farmworker families.

DETAILED DESCRIPTION:
This is a continuation of a community-based participatory research program focusing on pesticide contamination in migrant farmworker communities. Oregon Health Sciences University's Center for Research on Occupational and Environmental Toxicology and the Oregon Child Development Coalition propose to extend the participatory research model that has been developed to increase community capacity and to build knowledge on the nature and extent of childhood exposures to pesticides and resulting health effects. The project includes involvement from representatives of academic institutions, child and family educational, health, and social services, and the agricultural community. We propose to extend our program of research beyond the state of Oregon to accomplish the following specific aims:

1. Develop and validate a pathway model of organophosphate pesticide exposure for children residing near tree fruit orchards,
2. Conduct a longitudinal investigation of pesticide residue analysis, work practices, home characteristics and biological markers of exposure in migrant families residing in multiple homes and communities throughout a year,
3. Evaluate specific neurobehavioral outcomes in Latino children who speak Spanish and indigenous languages, living in homes with measured pesticide residues and in children living in homes with minimal measurable pesticide residues, and
4. Assess effectiveness of accepted methods of intervention including health education and environmental exposure reduction on changing behavior and reducing pesticide exposure in the migrant agricultural community.

The project also includes mechanisms to strengthen and expand the partnerships among migrant farmworker communities to increase the capacity of the community to address issues of environmental exposures and health. Training opportunities are provided for youth from the Latino farmworker community in environmental issues in affected communities. In addition to measuring the outcome of our research interventions in modifying exposures to pesticides and resulting health effects we have incorporated a comprehensive evaluation plan including measures to document increased research capacity in the community, leveraging by obtaining additional funding for further efforts, sustainability, culturally appropriate tools, policy or systems change, and impact on the field.

ELIGIBILITY:
Working in agriculture.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2000-07; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States